CLINICAL TRIAL: NCT05246176
Title: Role of Ultrasonography as a Single Tool for Guidance of Percutaneous Transhepatic Biliary Drainage in Obstructive Jaundice
Brief Title: Ultrasonography as a Single Tool for Guided Percutaneous Transhepatic Biliary Drainage in Obstructive Jaundice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Aboelmakarem Ahmed, Principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-22-1-02
Record Dates: First submitted 2022-01-12; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Jaundice
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental): group of patient with inoperable malignant obstructive jaundice with failed internal drainage.
  Interventions: Device: nephrostomy set

INTERVENTIONS:
Device: nephrostomy set — insertion of the nephrostomy set through the skin to obtaining good external drainage of bile in case of malignant obstructive jaundice.

SUMMARY:
Obstructive jaundice may be of malignant and benign etiologies. Carcinoma of the gall bladder, cholangiocarcinoma, pancreatic adenocarcinoma, metastasis, and lymph nodal compression of common bile duct (CBD) constitute the majority of malignant causes.

Most of the patients with malignant obstructive jaundice are already advanced and inoperable by the time they are diagnosed, hence carry bad prognosis with palliation being the only option left. Obstruction needs to be drained even in such cases for reducing pain, cholangitis, anorexia and pruritus as well as to reduce the serum bilirubin levels in certain cases to initiate chemo or intrabiliary brachytherapy.

Over the years, palliation has evolved with the introduction of newer methods and improvisation of existing techniques. Recent palliative measures prolong longevity and improve the quality of life, hence increasing the acceptance to such procedures; Methods of biliary drainage include: a. Surgical bypass b. Minimally invasive procedures; Endoscopic retrograde (ERCP) (cholangiopancreatography (ERCP), and Percutaneous transhepatic biliary drainage (PTBD).

ERCP as well as PTBD are well-established and effective means for biliary drainage as palliative treatment in unresectable cases.

With the current modern technique in experienced hands, Percutaneous Transhepatic Biliary Drainage (PTBD) equals endoscopic retrograde cholangio pancreatography (ERCP) regarding technical success and complications. In addition, there is a reduction in immediate procedure-related mortality with proven survival benefit. Moreover, it is the only immediate lifesaving procedure in cholangitis and sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Any adult Patients with malignant obstructive jaundice will included in this study

Exclusion Criteria:

* Patients with bleeding diathesis.
* Patients with associating comorbidities.
* Patients with insufficient intrahepatic biliary dilatation < 0.5 cm or with extensive tumor infiltrates.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Correction of hyperbilirubinemia. | 4 weeks
  We correct hyperbilirubinemia in patient with malignant obstructive jaundice using ultrasound to insert external drain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Venkatanarasimha N, Damodharan K, Gogna A, Leong S, Too CW, Patel A, Tay KH, Tan BS, Lo R, Irani F. Diagnosis and Management of Complications from Percutaneous Biliary Tract Interventions. Radiographics. 2017 Mar-Apr;37(2):665-680. doi: 10.1148/rg.2017160159. PMID 28287940
- [Background] Yarmohammadi H, Covey AM. Percutaneous biliary interventions and complications in malignant bile duct obstruction. Chin Clin Oncol. 2016 Oct;5(5):68. doi: 10.21037/cco.2016.10.07. PMID 27829281
- [Background] Gamanagatti S, Singh T, Sharma R, Srivastava DN, Dash NR, Garg PK. Unilobar Versus Bilobar Biliary Drainage: Effect on Quality of Life and Bilirubin Level Reduction. Indian J Palliat Care. 2016 Jan-Mar;22(1):50-62. doi: 10.4103/0973-1075.173958. PMID 26962281